CLINICAL TRIAL: NCT00724061
Title: Pilot Study of Pegylated Interferon-Alfa 2b in Combination With PUVA Therapy in Cutaneous T-Cell Lymphoma
Brief Title: Study of Pegylated Interferon-Alfa 2b in Combination With PUVA Therapy In CTCL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed early due to poor accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 07H4; P30CA060553 (NIH); NU 07H4 (Other: Northwestern University); SPRI-NU-07H4; STU00002993 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-07-26; First posted 2008-07-29 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2013-11

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — peginterferon alfa-2b; Furocoumarins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-IFN-α-2b + UV therapy (Experimental): Pegylated interferon α-2b in combination with UV therapy (either PUVA or NB-UVB).
  Interventions: Biological: Pegylated interferon α-2b; Other: Psoralens with ultraviolet light A; Other: Narrowband-ultraviolet light B

INTERVENTIONS:
Biological: Pegylated interferon α-2b — PEG-IFN-α-2b will be administered subcutaneously once a week. The starting dose of PEG-IFN-α-2b will be 1.5μg/kg. Each patient will undergo dose escalation to 3, 4.5, 6, 7.5, and up to 9μg/kg every 2 weeks or to maximum tolerated dose will be allowed. If no dose limiting toxicity (DLT) is observed, the maximum dose reached will be expanded. Once this dose has been given weekly for 2 weeks with no DLT, therapy will continue at this dose for up to 1 year depending on response.
  Other Names: PEG-Interferon alfa-2b; PEG-IFN-α-2b; PEG-Intron
Other: Psoralens with ultraviolet light A — Oral psoralen (8-methoxypsoralen, 0.6-1.0 mg/kg) will be taken 1.5 to 2 hours prior to UVA treatment. The initial UVA dosage will be approximately 0.5 to 1.5 J/cm2, and will be increased in increments as determined by skin type and tolerability. PUVA therapy will be given 2-3 times per week until complete remission (CR) is achieved. Afterwards, additional maintenance therapy will be given with a gradual reduction from once a week to every 4-6 weeks up to 1 year after CR was achieved.
  Other Names: PUVA
Other: Narrowband-ultraviolet light B — The initial NB-UVB dose will be 70% of the patient's MED and approximately 0.2 J/cm2 and will be increased by 15% of each subsequent treatment as determined by skin type and/or tolerability. Therapy will be given 3 times per week until complete remission (CR) is achieved. Additional maintenance therapy will be administered while gradually reducing NB-UVB from thrice weekly to once a week. All patients will continue maintenance NB-UVB therapy until 1 year after they have achieved CR.
  Other Names: NB-UVB

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may interfere with the growth of cancer cells and slow the growth of mycosis fungoides/Sezary syndrome. Ultraviolet light therapy uses a drug, such as psoralen, that is absorbed by cancer cells. The drug becomes active when it is exposed to ultraviolet light. When the drug is active, cancer cells are killed. Giving PEG-interferon alfa-2b together with ultraviolet light therapy may kill more cancer cell.

PURPOSE: This is a pilot study of dose-escalating pegylated IFN-α-2b and PUVA or NB-UVB. The purpose is to study the side effects and best dose of PEG-interferon alfa-2b to be given together with ultraviolet light therapy in patients with stage IB, stage II, stage III, or stage IVA mycosis fungoides/Sezary syndrome (CTCL).

DETAILED DESCRIPTION:
Patients receive PEG-interferon alfa-2b subcutaneously once weekly for 12 months in the absence of disease progression or unacceptable toxicity. Patients also receive UV light therapy (either PUVA or NB-UVB).

Health-related quality of life is assessed periodically using the FACT-BRM, FACT-G, and FACT-CTCL questionnaires.

After completion of study therapy, patients are followed for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mycosis fungoides/Sezary syndrome

  * Stage IB-IVA disease
  * Erythrodermic disease allowed
* Measurable disease

  * One or more indicatory lesions must be designated prior to study entry

PATIENT CHARACTERISTICS:

* ECOG/WHO performance status 0-1
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* WBC ≥ 3,000/mm³
* Serum creatinine ≤ 2.0 mg/dL
* Total serum bilirubin ≤ 2.2 mg/dL
* Serum AST and ALT ≤ 2 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients must be disease free of prior malignancies for ≥ 5 years except currently treated squamous cell or basal cell carcinoma of the skin, carcinoma in situ of the cervix, or surgically removed melanoma in situ of the skin (stage 0), with histologically confirmed free margins of excision
* No history of seizure disorder or severe heart disease
* No acute infections
* Diagnosed depression allowed with receiving appropriate care for depression

PRIOR CONCURRENT THERAPY:

* No prior psoralens with ultraviolet light A or interferon alfa therapy
* More than 4 weeks since prior topical therapy, systemic chemotherapy, or biologic therapy
* More than 4 weeks since prior surgery and fully recovered
* At least 1 week since prior antibiotics
* No other concurrent standard or investigational topical and systemic antipsoriatic or anticancer therapies including radiation, steroids, retinoids, nitrogen mustard, thalidomide, or other investigational agents
* No concurrent topical agents except emollients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened at Northwestern University in 09/2008 with an accrual goal of 15 subjects. The study was suspended from 11/2009 to 07/2010 due to a shortage of psoralens; a revision allowed the use of PUVA or NB-UVB for UV therapy.
  A total of 7 patients were enrolled before the study was closed due to poor accrual in 05/2012.
Groups:
- PEG-IFN-alpha-2b + UV Therapy: Pegylated interferon α-2b in combination with UV therapy (either PUVA or NB-UVB).
Period: Dose Escalation Phase
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Started | 7
Completed | 2
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Disease Progression | 3
Period: Maintenance Therapy
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Number analyzed (Participants) | 7
Age, Customized [Number; unit: participants]
  30-39 | 1
  40-49 | 2
  50-59 | 2
  60-69 | 0
  70-79 | 2
  80-89 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) Observed During Dose Escalation of PEG-IFN-α-2b
Description: Adverse events are graded according to the National Cancer Institute's Common Toxicity Criteria (CTCAE) version 3.0. In general, grades are assigned as follows:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
  A dose limiting toxicity (DLT) will be defined as any grade 3 or higher hematologic toxicity or any grade 4 non-hematologic toxicity.
Time Frame: From the date that the first patient began treatment until the last patient completed the dose escalation phase (up to 12 weeks per patient)
Measure: Number; unit: dose limiting toxicities
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Number analyzed (Participants) | 7
dose limiting toxicities | 0

2. Primary Outcome: Change in Total Health-related Quality of Life Score Using the Functional Assessment of Cancer Therapy - Biologic Response Modifier (FACT-BRM)
Description: The FACT-BRM is a patient self-report tool to assess health-related quality of life measures.
Time Frame: During 12 weeks of dose escalation and then up to one year during maintenance therapy.
Population: No data collected for this outcome measure.
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients Exhibiting a Complete Response
Description: Response was assessed according to the Composite Assessment of Index Lesion Disease Severity. Clinical signs are graded on scales of 0 to 8 (0 being no evidence of disease and 8 being the near worst severity of sign/symptom). The CA response is calculated as the ratio of the sum of the grades for all clinical signs plus the surface areas for all index lesions at each visit compared to the sum of these grades at baseline. The CA also considers all other cutaneous lesions and any extra-cutaneous manifestations of disease.
  CR requires a CA ratio of 0 (zero) with no evidence of new disease (abnormal or pathologically positive lymph nodes, cutaneous or other tumor manifestations, visceral disease) present over 4 weeks. Patients with Sézary Syndrome must have no evidence of circulating Sézary cells (< 5% Sézary cells are considered to be not significant). Skin biopsy is required for documentation of CR.
Time Frame: During 12 weeks of dose escalation and then up to one year during maintenance therapy.
Population: No data collected for this outcome measure.
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: To Evaluate the Duration of Response
Description: To evaluate duration of response related to combined pegylated IFN-α-2b plus PUVA or NB-UVB therapy.
Time Frame: At each study visit
Population: No data collected for this outcome measure.
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in Activation Status of Key Signaling Molecules Between Baseline and After 2 Weeks of Treatment
Description: The activation status of key signaling molecules affecting the PI3K and JAK/STAT pathways was to be analyzed in samples of skin and blood taken at baseline and after 2 weeks of treatment. Participation in this exploratory component of the trial was optional for patients.
Time Frame: At baseline and after 2 weeks of treatment (for those patients who consented to this portion)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Correlation of Response With Infiltration of Skin Lesions With Dendritic Cells, Cytotoxic CD8+ T-cells, and NK-cells
Time Frame: Baseline, 24 hours post-1st dose in the dose escalation phase, and 24 hours post-1st dose in the maintenance therapy phase
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date the first patient began treatment until 30 days after the last patient went off study treatment.
Arm/Group | PEG-IFN-alpha-2b + UV Therapy
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN-alpha-2b + UV Therapy (N=7)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1) — Pain and/or swelling with inflammation or phlebitis
Ventricular arrhythmia - ventricular tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN-alpha-2b + UV Therapy (N=7)
ALT, SGPT elevation (Metabolism and nutrition disorders) | 4 (5)
AST, SGOT elevation (Metabolism and nutrition disorders) | 5 (6)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (7)
Anorexia (Gastrointestinal disorders) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 1 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Constitutional symptoms - other (fever, chills, sweats, aches & pains) (General disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine - elevation (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 6 (7)
Fever (General disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (7)
Hemoglobin (decrease) (Blood and lymphatic system disorders) | 4 (5)
Hypopigmentation - slight or localized (Skin and subcutaneous tissue disorders) | 1 (1)
Infection - skin (cellulitis) (Skin and subcutaneous tissue disorders) | 1 (2)
Insomnia (General disorders) | 1 (2)
Leukocytes (total WBC) - decreased (Blood and lymphatic system disorders) | 5 (8)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6)
Musculoskeletal/soft tissue - other (injection site pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) - decreased (Blood and lymphatic system disorders) | 3 (7)
Odor (patient) (General disorders) | 1 (1)
Other impact on blood/bone marrow (Blood and lymphatic system disorders) | 2 (2)
Pain - head/headache (General disorders) | 3 (4)
Pain - muskuloskeletal (Musculoskeletal and connective tissue disorders) | 2 (3)
Platelets (decreased) (Blood and lymphatic system disorders) | 3 (6)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Pruritus/itching - mild or localized (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Weight loss - intervention not indicated (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Only 7 patients were enrolled before the study was terminated by the Data Monitoring Committee due to poor accrual. Accrual was limited by a worldwide psoralen shortage and well as the exclusion of patients with prior UV light exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes